CLINICAL TRIAL: NCT04567407
Title: Bilateral Continuous Erector Spinae Blocks for Post-Sternotomy Pain Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Roland Brusseau, Director of Regional Anesthesia Program, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00034302
Record Dates: First submitted 2020-09-18; First posted 2020-09-28 (Actual); Results first posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Pain
Keywords: regional anesthesia; cardiac surgery; erector spinae
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Prospective single-arm intervention trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bilateral erector spinae blocks (Experimental): All enrolled patients will have bilateral erector spinae blocks (with catheters for postoperative local anesthetic infusion) placed by the by a member of the clinical regional anesthesia team (under the supervision of a member of the research team) in a sterile fashion after the cardiac surgical procedure is completed. Postoperative continuous infusion of local anesthetic (ropivacaine) via the nerve block catheter is initiated and managed by the Acute Pain Service (per standardized, clinical weight-based protocols).
  Interventions: Drug: Bilateral erector spinae blocks using ropivacaine

INTERVENTIONS:
Drug: Bilateral erector spinae blocks using ropivacaine — Bilateral chest wall nerve blocks using ropivacaine.
  Other Names: Naropin

SUMMARY:
To evaluate the efficacy of bilateral continuous erector spinae blocks (BESB) for postoperative analgesia in children and adolescents undergoing cardiac surgical procedures via sternotomy in the Early Recovery After Surgery (ERAS) program in a single arm, open label, interventional study.

DETAILED DESCRIPTION:
Regional anesthesia-and pediatric regional anesthesia in particular-is a rapidly evolving subfield of anesthesia practice driven with considerable urgency by the growing recognition that even appropriate perioperative opioid administration can have significant deleterious long-term effects.

Regional anesthetics can provide targeted, continuous analgesia to select dermatomes with minimal additional patient risk and as such, have become routine components of opioid-sparing intraoperative and postoperative pain management plans for non-cardiac surgical patients at a single institution. In addition to the postulated benefit of reducing overall opioid exposure (and potentially reducing the risk for long term physiologic and behavioral dependence upon opioids), regional anesthetics may allow for earlier extubation after selected surgeries, shorter intensive care unit (ICU) stays, shorter inpatient admissions, earlier mobilization, fewer gastrointestinal complications, and improved patient and care team satisfaction scores.

Historically, regional anesthetics have been avoided in cardiac surgery as most patients are pharmacologically anticoagulated during their procedures and are thus at increased risk for bleeding. This is particularly worrisome in the pediatric cardiac surgical population as many of these children remain intubated for an extended period of time postoperatively and therefore may not have reliable neurological exams in the setting of neuraxial regional anesthetics-potentially resulting in unrecognized hemorrhage-related acquired neurological deficits.

Recently, the erector spinae block (ESB) has become popular for providing analgesia after a number of anterior chest and abdominal procedures. This simple interfascial plane block can reliably provide unilateral chest and/or abdominal wall analgesia. It has been described in numerous case reports and case series as an effective block for management of unilateral thoracotomies, unilateral rib fractures, unilateral abdominal incisions and most notably, for management of post-sternotomy pain when applied bilaterally. New case reports and series involving the ESB are being published almost weekly with a growing number of manuscripts specific to cardiac surgical applications. Indeed, numerous randomized controlled trials have investigated the analgesic efficacy of bilateral erector spinae plane blocks (BESB) compared with conventional treatment for pain after cardiac surgery in adult patients and have been published recently (2018-2019) with promising results.

As an interfascial plane block in a compressible anatomical space, the ESB is considered safe in anticoagulated (or recently anticoagulated) patients. It is fast becoming a preferred anesthetic option at BCH for anticoagulated patients - as opposed to neuraxial (e.g. epidural) and paraneuraxial blocks (i.e. paravertebral) nerve blocks, which are largely contraindicated in this setting. Further, given its relative ease of placement, apparent efficacy and safety profile, it is increasingly becoming a standard option for patients undergoing a wide range of thoracic, abdominal and thoraco-abdominal procedures.

The investigators recently investigated the feasibility of performing these blocks bilaterally in a pediatric cardiac surgical population undergoing sternotomy-based procedures (IRB-P00031524). At the conclusion of this 10-patient pilot, the investigators found that performing these blocks was technically feasible, requiring 30 minutes or less of OR time, resulting in no known complications. Furthermore, the data suggested an approximate 25% reduction in rescue opioid requirements in the first 48 hours amongst the erector spinae group (p=0.048).

In order to best evaluate the efficacy of this block in the pediatric cardiac population, a blinded, randomized and controlled trial would be ideal. However, given that randomization could be challenging and the fact that blinding would not be feasible, the investigators believe an observational prospective cohort study is most appropriate at this time.

As such, the investigators propose to evaluate the comparative efficacy of BESB versus matched historical controls who received standard of care pain management (systemic opioid therapy) for patients undergoing cardiac surgery via sternotomy by means of a single arm, open label, interventional study that will compare as the primary outcome rescue analgesic requirements, rendered as opiate equivalents, at 12, 24 and 48 hours, and the 24 hour period preceding both 72 and 96 hours postoperatively. 'Efficacy' will be considered as a threshold of clinical significance being defined as a 15% difference). In addition to the primary endpoint, we plan to evaluate the duration of intubation, length of ICU stay, median pain scores, incidence of PONV (postoperative nausea and vomiting; 0-6h, 6-12h and overall), time to mobilization and adverse events between these groups. Postoperative data collected from standard clinical follow-up tools, such as return to baseline sleep and activity status as well as pain medication requirements at home, will also be compared. In addition, the investigators plan to evaluate the quality of sleep and activity with a smart watch (Fitbit™ ) during the perioperative period in the BESB group only.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled as part of the cardiac surgical ERAS program: Patients scheduled for elective surgeries for the following congenital anomalies, or similar: atrial septal defects (all types), partial anomalous pulmonary venous connection (non-obstructed), cor-triatriatum, VSD, partial AV canal, sub-aortic membrane resection, anomalous aortic origin of the coronary arteries, and pulmonary valve/conduit implantation
2. Scheduled for a primary sternotomy.
3. Ages 2 years through 17 years.

Exclusion Criteria:

1. Single ventricle physiology.
2. Significant scoliosis or other anatomic contraindications to ESB.
3. Significant intraoperative hemodynamic instability or bleeding, as ascertained by clinicians taking care of the patient.
4. Patients with severe neurodevelopmental delays.
5. Patients with previous chronic pain syndromes.
6. Patients with a history of greater than 24 hours of postoperative or post-procedural opioid treatment at any point in the 2 months prior to surgery.
7. Lack of parental consent and/or child assent.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2022-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ROLAND BRUSSEAU, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children"S Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bilateral Erector Spinae Blocks
Started | 45
Completed | 40
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Bilateral Erector Spinae Blocks
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 45
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 11.15 [5.17 to 15.15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Analgesic Requirement
Description: Total opiate equivalents
Time Frame: 24hours postop
Measure: Mean (Standard Error); unit: (mg/kg)
Arm/Group | Bilateral Erector Spinae Blocks
Number analyzed (Participants) | 40
(mg/kg) | 0.60 (0.06)

2. Primary Outcome: Analgesic Requirement
Description: Total opiate equivalents
Time Frame: 48hours postop
Measure: Mean (Standard Error); unit: mg/kg
Arm/Group | Bilateral Erector Spinae Blocks
Number analyzed (Participants) | 40
mg/kg | 1.13 (0.08)

3. Primary Outcome: Analgesic Requirement
Description: Total opiate equivalents
Time Frame: 96hours postop
Measure: Median (Inter-Quartile Range); unit: (mg/kg)
Arm/Group | Bilateral Erector Spinae Blocks
Number analyzed (Participants) | 40
(mg/kg) | 1.34 [0.87 to 2.00]

4. Secondary Outcome: Duration of Mechanical Ventilation/Intubation
Description: Length of postoperative mechanical ventilation/intubation following OR exit
Time Frame: 48hrs
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Bilateral Erector Spinae Blocks
Number analyzed (Participants) | 40
hours | 0.7 [0 to 6.0]

5. Secondary Outcome: Length of Postoperative ICU Stay
Description: Duration of ICU stay following OR exit
Time Frame: 72Hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Bilateral Erector Spinae Blocks
Number analyzed (Participants) | 40
hours | 23.3 [22.1 to 50.1]

6. Secondary Outcome: Length of Hospital Stay
Description: Duration of Inpatient hospital admission
Time Frame: 5 Days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Bilateral Erector Spinae Blocks
Number analyzed (Participants) | 40
days | 4.10 [3.83 to 5.08]

7. Secondary Outcome: Median Pain Scores
Description: Patient reported pain scores using either NRS score (numeric rating scale of 1-10, with 10 being the worst pain), the INRS score (individualized numeric rating scale of 1-10, with 10 being the worst pain) or FLACC scale (face, legs, activity, cry, consolability scale of 0-10 with 10 being the worst pain). Patients were assessed multiple times (variably - per routine clinical practice, every few hours during the Time Frame) in order to derive a median for each participant per 12h period. Median pain scores were used rather than time specific pain scores to compare patients in the single arm cohort study to controls from the ERAS controls. Median pain scores were averaged across all participants in the intervention arm as well as the controls. Outcomes are reported as mean with the standard error.
Time Frame: day of surgery (POD 0) 7:00am - 18:59pm
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Bilateral Erector Spinae Blocks
Number analyzed (Participants) | 40
score on a scale | 3.30 (0.59)

8. Secondary Outcome: Median Pain Scores
Description: as for outcome 7
Time Frame: night of surgery (PON 0) 19:00pm-6:59am
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Bilateral Erector Spinae Blocks
Number analyzed (Participants) | 40
score on a scale | 3.46 (0.04)

9. Secondary Outcome: Median Pain Scores
Description: as for outcome 7
Time Frame: Post-Op Day 1 (7:00am-18:59pm)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Bilateral Erector Spinae Blocks
Number analyzed (Participants) | 40
score on a scale | 3.18 (0.30)

10. Secondary Outcome: Median Pain Scores
Description: as for outcome 7
Time Frame: Post-Op Night 1 (19:00pm-6:59am)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Bilateral Erector Spinae Blocks
Number analyzed (Participants) | 40
score on a scale | 2.92 (0.33)

11. Secondary Outcome: Time to First Mobilization
Description: Time to out of bed activity (e.g., up to chair, ambulation)
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Bilateral Erector Spinae Blocks
Number analyzed (Participants) | 40
hours | 6.75 [5.03 to 9.83]

ADVERSE EVENTS:
Time Frame: 30 days
Description: All patients were rounded on by study team members daily while in hospital. Per routine standard of care, they saw a Physician Assistant on POD 7 with a standardized questionnaire, they received patient reported outcomes surveys at 5, 10 and 20 days and they had a virtual 30-day questionnaire. In addition, all additional postoperative visits were reviewed, including Emergency Department admissions, as applicable.
Arm/Group | Bilateral Erector Spinae Blocks
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 10/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bilateral Erector Spinae Blocks (N=40)
Catheter obstruction - unilateral (Skin and subcutaneous tissue disorders) | 2 (2)
Catheter leakage under dressing (Skin and subcutaneous tissue disorders) | 5 (5)
Bleeding/hematoma (Skin and subcutaneous tissue disorders) | 2 (2)
Chest wall paresthesia (Nervous system disorders) | 1 (1) — Unilateral chest wall paresthesia not following specific dermatome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT04567407/Prot_SAP_000.pdf